CLINICAL TRIAL: NCT06154785
Title: Low Stable Pressure Pneumoperitoneum in Colorectal Surgery : An Ideal Stage 2b Prospective International Cohort Study (CROSS STUDY)
Brief Title: Low Stable Pressure Pneumoperitoneum in Colorectal Surgery (CROSS STUDY)
Acronym: CROSS
Status: Recruiting | Type: Observational
Sponsor: Bordeaux Colorectal Institute Academy (Other)
Responsible Party: Sponsor
Other Study IDs: B.C.I.A 2023/01
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Surgery; Benign or Malignant Rectal or Colon Tumors
Keywords: colorectal pathology; low stable pressure; laparoscopic; length hospital stay
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- International cohort: This is an international cohort (France and other international centers) which consists of including patients undergoing colorectal surgery performed at low pressure for benign or malignant pathology.This stage 2b cohort study is a pilot study assessing the best operative association with stable low-pressure pneumoperitoneum in order to optimize postoperative outcomes after mini invasive colorectal surgery.

SUMMARY:
The objective of this prospective, international cohort is to incorporate the low stable pressure (using Airseal Insufflator) approach and its associated parameters into the early rehabilitation program after colorectal surgery so as to shorten hospitalization up to the ambulatory care and reduce postoperative pain and opioid consumption.

DETAILED DESCRIPTION:
Laparoscopy is currently the gold standard for the vast majority of abdominal surgeries, and especially for colectomy for cancer or benign diseases. There are many data showing the benefits of the laparoscopic approach to colectomy in terms of morbidity, post-operative pain and analgesic consumption, length of hospital stay, cosmetic results, and improved patient satisfaction. In 2002, consensus European guidelines recommended insufflating at the lowest pressure that still provides sufficient exposure. Considering these results, low-pressure laparoscopy is one of the alternatives that have been developed to do away with the complications of the pneumoperitoneum while retaining its advantages.

However, other factors may influence the outcomes of the low-pressure pneumoperitoneum such as the use of humidification and warming gaz, robotic or microsurgical instrumentation, neuromuscular blockade, patient positioning, pre-stretching of the abdominal wall, ventilation-induced changes, and probably individual patient factors like obesity. These parameters could not be separately tested in randomized trial. We should consider all these parameters in a prospective international registry in order to optimize the benefit of low-pressure pneumoperitoneum in post-operative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Colonic resection (right or left, subtotal or total) performed for benign or malignant pathology
* Rectal resection with or without stoma for benign or malignant pathology
* Laparoscopic or robotic procedure
* Surgery under low stable pressure pneumoperitoneum with AirSeal
* Patient who benefits by medicare system
* Oral agreement after reading information letter

Exclusion Criteria:

* Laparotomy procedure
* Associated resection (except appendectomy or liver biopsy)
* Transverse colectomy
* Emergency procedure
* Pelvic sepsis
* Pregnancy or breast feeding period
* Legal incapacity or physical, psychological social or geographical status interfering with the patient's ability to agree to participate in the study
* Persons deprived of liberty or under guardianship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This cohort study is a pilot study assessing the best operative association with stable low-pressure pneumoperitoneum in order to optimize postoperative outcomes after mini-invasive colorectal surgery. The use of robotic or microsurgical instrumentation, neuromuscular blockade, patient positioning, pre-stretching of the abdominal wall and ventilation-parameters could not be separately tested in randomized trial.
  In this pilot study, we aim to include 300 patients with low stable pneumoperitoneum with Colorectal surgery.
  All patient assessements will be done according to the sites standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
To assess the impact of the stable low-pressure approach (using Airseal Insufflator) and its associated parameters into the the early rehabilitation program after colorectal surgery on length of stay. | From the surgery to the end of the hospitalization (max 30 days)
  Evaluate the Length of hospital stay after colorectal surgery.

SECONDARY OUTCOMES:
The impact of stable low pressure on the postoperative pain after colorectal surgery | At 24 hours after the end of the surgery
  Pain is evaluated (Visual Analgesic Scale (Vas scores from 0 (no pain) to 10 (hurst worst))
The impact of stable low pressure on the opioid consumption after colorectal surgery | From the surgery to the end of the hospitalization (max 30 days)
  Evaluate the impact on the opioid consumption after colorectal surgery;
The impact of the different mini-invasive approaches on the feasibility and benefit of low stable pressure | From the surgery to the end of the hospitalization (max 30 days)
  Evaluate the impact of robotic, laparoscopic +/- microsurgical instrument, 3D laparoscopic vision surgery
The Post-operative Surgical and Medical morbidity | From the surgery to the end of the hospitalization (max 30 days)
  Post operative Surgical and Medical morbidity according to the Clavien-Dindo Classification
The impact of the anesthetic management on the feasibility and benefit of low stable pressure | From the surgery to the end of the hospitalization (max 30 days)
  Evaluate the impact of drugs, deep neuromuscular blockade, ventilation characteristics, intraoperative nociception monitoring, patient positioning, pre-stretching of the abdominal wall, and individual patient factors
The Surgical and Medical morbidity at 30 days | At 30 days after the end of the surgery
  Surgical and Medical morbidity at 30 days according to the Clavien-Dindo Classification

CONTACTS AND LOCATIONS:
Locations (18):
- Universitair Ziekenhuis, Jette, Brussels Capital, Belgium
- France (11):
  - Hôpital Jean Minoz, Besançon
  - Clinique Tivoli-Ducos - Bordeaux Colorectal Institute, Bordeaux
  - Hôpital Albert Michallon, La Tronche
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Nord-Marseille, Marseille
  - Clinique Hartmann, Neuilly-sur-Seine
  - Hopital Saint-Louis, Paris
  - Hôpital Saint-Antoine, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Lyon Sud, Pierre-Bénite
  - Hopital Charles Nicolle, Rouen
- St. Georg Klinikum Eisenach, Eisenach, Germany
- Division of Colon and Rectal Surgery, Milan, Italy
- Academic Medical Center, Amsterdam, Netherlands
- Hospital General Universitario Gregorio, Madrid, Spain
- Hôpitaux Universitaires de Genève, Geneva, Switzerland
- Nhs Fundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data (IPD) with other researchers